CLINICAL TRIAL: NCT07243535
Title: Comparison Between a Session of Walking Synchronized to Fractal- VS Isochronous-Based Cues on Gait Variability and Corticospinal Measures in Athletes With a Reconstructed Anterior Cruciate Ligament: A Crossover Randomized Controlled Trial
Brief Title: Fractal vs Isochronous Cueing in Athletes After ACL Reconstruction
Acronym: SyncGait
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SyncGait-5725
Record Dates: First submitted 2025-09-16; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Anterior Cruciate Ligament Reconstruction; Anterior Cruciate Ligament Reconstruction Rehabilitation; Athlete
Keywords: Complexity; Excitability; Metronome; Neuroplasticity; Rehabilitation

STUDY DESIGN:
Intervention Model Description: This study is a crossover randomized controlled trial, comprising two sessions. Each session will take approximately 2 hours, and the sessions will be separated from 7 to 10 days. Both sessions will be held at the same period of the day to avoid the circadian effect on our primary outcome. The two sessions will be similar. At the beginning of the first session, however, three questionnaires will be administered to collect the demographic and baseline characteristics of the participants. Following the completion of these questionnaires, a randomization process through a fixed block method will be conducted by the study's supervisor to determine the order in which the intervention will be presented across the two sessions. The participants will be asked to complete three 12-minute gait trials in each session: one cued trial and two uncued trials. A minimum of 20 minutes of rest will be taken between each trial while collecting the cortical drive assessment, PRE and POST the cued trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: The randomized order will be transmitted only to the main researcher through a sealed envelope. Participants will be blinded throughout their participation. Importantly, the participants are unable to detect the subtle changes in variability between the Isochronous and Fractal cueing conditions. The main researcher will not be blinded for the condition given the necessity to program the metronome per session. However, the remaining team will be blinded and, therefore, will run the data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fractal Cueing, Then Isochronous Cueing (Experimental): Participants exposed to 12-minute treadmill walking synchronized to a visual fractal metronome individualized to stride time variability. After a washout period of 1 week, participants will be exposed to 12-minute treadmill walking synchronized to a visual isochronous metronome with fixed stride time.
  Interventions: Device: Fractal Cueing; Device: Isochronous Cueing
- Isochronous Cueing, then Fractal cueing (Experimental): Participants exposed to 12-minute treadmill walking synchronized to a visual isochronous metronome with fixed stride time. After a washout period of 1 week, participants will be exposed to 12-minute treadmill walking synchronized to a visual fractal metronome individualized to stride time variability.
  Interventions: Device: Fractal Cueing; Device: Isochronous Cueing

INTERVENTIONS:
Device: Fractal Cueing — Walking synchronized to a visual fractal metronome.
Device: Isochronous Cueing — Walking synchronized to a visual Isochronous metronome.

SUMMARY:
Anterior cruciate ligament (ACL) injuries are among the most prevalent and functionally limiting knee injuries in sports, particularly those that involve pivoting movements. Despite advancements in surgical reconstruction and physical rehabilitation, many athletes continue to exhibit persistent motor control deficits and increased gait variability, both of which are closely linked to a heightened risk of re-injury and long-term joint degeneration. These deficits arise from biomechanical impairments and disrupt proprioceptive input that requires cortical reorganization, contributing to maladaptive neuroplasticity. However, conventional rehabilitation strategies often overlook this neural dimension. Recent findings emphasize the importance of fostering motor variability and promoting neuroplasticity through external focus strategies, including sensorimotor synchronization. While isochronous cues, an invariant stimulus, are commonly used, they do not reflect the natural fluctuations of healthy gait and may reduce its complexity. Fractal-based cues, in contrast, introduce structured variability resembling the natural dynamics of locomotion and have been shown to restore gait complexity in clinical populations. However, no study has yet explored their acute effects on gait variability and corticospinal function following ACL reconstruction (ACLR). This crossover randomized controlled trial aims to compare the acute effects of a single session of treadmill walking synchronized to either fractal or isochronous-based visual cues on gait variability and corticospinal measures in athletes with ACLR. The investigators hypothesize that fractal-based cueing will acutely restore gait variability and enhance corticospinal excitability, evidenced by increased corticospinal excitability and intracortical facilitation, and reduced short-interval intracortical inhibition, thus promoting adaptive neuroplasticity. Conversely, isochronous cueing is expected to maintain or decrease gait complexity without improving corticospinal measures. This study may provide insights that could be highly valuable as a way to promote neuroplasticity and optimize gait rehabilitation after ACLR, also allowing an objective quantification and aiming to restore variability to levels close to those observed in healthy individuals, thus contributing to reducing the re-injury rate.

DETAILED DESCRIPTION:
This study will test a laboratory-based intervention using gait trials with sensorimotor synchronization, a common approach in gait rehabilitation aimed at restoring or acutely modifying gait variability. The intervention, called SyncGait, consists of treadmill walking synchronized with visual cues. Following a crossover design, each participant will complete two sessions, one with fractal cueing (FRC) and one with isochronous cueing (ISO), with the order randomized. Each cued trial will last 12 minutes and will be preceded and followed by uncued walking trials. The visual cues will be presented as a moving bar on a screen positioned in front of the treadmill. For the FRC condition, the cues will be individualized to each participant's stride time variability, generated through a fractal algorithm and validated using detrended fluctuation analysis. For the ISO condition, cues will match each participant's average stride time without variability. Participants will be instructed to synchronize heel strikes of the reconstructed limb with the top of the moving bar. The treadmill (Bertec Inc., USA) will record gait data at 1000 Hz. Each session will be conducted individually, supervised by at least two trained team members. A sample size of 36 participants was determined to ensure adequate power (90%) to detect a moderate effect size (ηp² = 0.25) at a 5% significance level, accounting for an anticipated 20% dropout rate. To encourage participation and retention, participants will receive a personalized evaluation report and a free isokinetic assessment within 12 months. Data collection will include both gait and corticospinal outcomes. Gait variability will be analyzed from treadmill force data, focusing on stride intervals and synchronization performance. Corticospinal outcomes will be assessed using transcranial magnetic stimulation (TMS) with a BiStim2 stimulator (Magstim®, UK). Electromyography (Delsys Trigno, AD Instruments, NZ) will be recorded from quadriceps and hamstrings, while knee strength will be assessed with an isokinetic dynamometer (Humac Norm, USA). Standardized electrode placement and contraction protocols will ensure reproducibility. During testing, single- and paired-pulse TMS protocols will be applied at 10% of maximal voluntary contraction. Ten stimuli per condition will be collected, providing reliable estimates of excitability and inhibition. Visual feedback will help participants maintain the required contraction level throughout assessments. Statistical analysis will begin with normality testing (Shapiro-Wilk). Linear mixed models (Time × Cue condition) will be used for primary and secondary outcomes. Post-hoc comparisons will use Bonferroni corrections. Synchronization accuracy will be compared with paired t-tests. Statistical significance will be set at p < 0.05, and analyses will be performed using Jamovi software. This protocol is designed to rigorously test whether fractal cueing can restore healthy gait variability patterns and enhance corticospinal excitability in athletes with ACL reconstruction, compared with conventional isochronous cueing.

ELIGIBILITY:
Inclusion Criteria:

* Undergone unilateral ACL reconstruction less than 2 years ago;
* Have medical release for the full load on the injury limb for at least 2 weeks;
* Be independently pain-free walking;
* Being sports athletes according to an athlete description: Training regularly to improve performance, actively participating in competitions or formally registering in a sports federation or association;
* Must be able to understand and perform the requested task.

Exclusion Criteria:

* Participants with previous surgery on either knee;
* Those with more than 3 months between ACL injury and surgery;
* More than 2 weeks between surgery and the start of physical therapy;
* Had another musculoskeletal injury in the lower limb within the past 6 months;
* Another musculoskeletal surgery within the past 18 months;
* Participants with a history of movement system pathologies, such as nervous system, cardiovascular, pulmonary, integumentary, or endocrine conditions;
* Participants with vestibular or somatosensory system pathologies or visual impairments limiting their ability to see the metronome required for the task;
* Use of medications that could affect locomotion and balance.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Gait Variability Measured by Fractal Scaling Exponent of inter-stride intervals | Pre- (40 minutes before) and Post- (40 minutes after) -Intervention
  The fractal-scaling exponent, α, of inter-stride intervals (α-ISIs) will be determine by calculating the time between two consecutive heel strikes of the same foot. First, the investigators will identify the heel strike events of the dominant foot. To improve the identification of this event, the signals will be filtered using a 2nd order, zero lag low-pass Butterworth filter with a cutoff frequency of 20 Hz. Then, Detrended Fluctuation Analysis (DFA) will be used to determine the fractal-scaling, an index of complexity. The DFA is a modified random-walk analysis that makes use of a long-range correlated time series. The long-range correlation can be mapped to self-similar calculations through simple integration.
Corticospinal Excitability Measured by Motor Evoked Potential Amplitude | Baseline (Pre) and immediately after the intervention (Post)
  Conducted using Spike2 software (version 10; Cambridge Electronic Design, Cambridge, United Kingdom) and subsequently exported to, MATLAB R2018a (The MathWorks, Natick, Massachusetts, United States) for processing and analysis. Corticospinal Excitability will be quantified as the peak-to-peak amplitude of MEPs elicited by a single-pulse TMS stimulus, with values averaged across 10 trials per participant.
Cortical Silent Period (SP) Duration | Baseline (Pre) and immediately after the intervention (Post)
  Silent period will be calculated as the time from MEP onset to the resumption of voluntary EMG activity, expressed as SP = resumption of voluntary EMG time - MEP onset (58), and averaged across all 10 stimuli.
Intracortical Facilitation (ICF) | Baseline (Pre) and immediately after the intervention (Post)
  ICF will be determined using the same calculation method but with an interstimulus interval of 12 ms (ICF = conditioned MEP / control MEP).
Short-Interval Intracortical Inhibition (SICI) | Baseline (Pre) and immediately after the intervention (Post)
  SICI will be calculated as the ratio between the conditioned MEP elicited with a paired-pulse TMS protocol (interstimulus interval: 3 ms) and a control MEP obtained from AMT assessment, expressed as SICI = conditioned MEP / control MEP.

SECONDARY OUTCOMES:
Magnitude of variability | Pre- (40 minutes before) and Post- (40 minutes after) -Intervention
  Calculate the coefficient of variation of inter-stride intervals, representing the magnitude of variability.
Synchronization Accuracy | During Intervention
  Asynchronies (ASYNC), i.e., the time difference between the heel strikes and the cues, expressed in milliseconds. This will be used to ensure that differences at the primary outcome are not the result of different synchronization performances. A negative value of ASYNC indicates that the heel strike occurred before the cue. The ASYNC provides information regarding the strategies used and the performance of the synching processes, serving as a control parameter to reliably interpret our results in terms of gait complex.

OTHER OUTCOMES:
Demographic characterization of the sample by Lysholm Knee Score (LKS). | At the beginning of the first session (Day 1)
  The LKS show good internal consistency (Cronbach's α = 0.802) and high test-retest reliability (ICC = 0.859). The LKS consists of 8 items with 3 to 6 closed-response options, assessing knee function aspects such as pain, swelling, locking, and instability. The scale is completed in ≈5 minutes, with higher scores indicating better knee function.
Demographic characterization of the sample by Tegner Activity Scale (TAS) | At the beginning of the first session (Day 1)
  The TAS show good internal consistency (Cronbach's α = 0.802) and high test-retest reliability (ICC = 0.972). The TAS comprises a single item with 11 activity levels (0-10), reflecting increasing physical demand. The scale is completed in ≈2 minutes, with higher scores indicating greater physical activity levels (TAS).
Demographic characterization of the sample by Tampa Scale of Kinesiophobia (TSK) | At the beginning of the first session (Day 1)
  The TSK consists of 13 items rated on a 4-point Likert scale (1 = strongly disagree to 4 = strongly agree), with a total score ranging from 13 to 52, where higher scores indicate greater kinesiophobia. It required 4 to 6 minutes to complete the instrument and demonstrated good internal consistency (α = 0.82) and test-retest reliability (ICC = 0.99), confirming its reliability for assessing kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: João R Vaz, PhD, Study Director — Egas Moniz school of Health & Science
Locations (1):
- Egas Moniz School of Health & Science, Almada, Monte de Caparica, Portugal

IPD SHARING:
Plan to Share IPD: Yes
All raw data will be stored in the supervisor's institutional personal Microsoft 365 account for five years, after which it will be permanently deleted. Data will be recorded anonymously using a unique coded numerical ID, known only to the supervisor. The database will be in Excel format. The encoded dataset may be shared with the rest of the research team and the journal where the study will be published, which may, in turn, make the data available to the scientific community for one year following publication.

REFERENCES:
- [Background] Grooms DR, Page SJ, Nichols-Larsen DS, Chaudhari AM, White SE, Onate JA. Neuroplasticity Associated With Anterior Cruciate Ligament Reconstruction. J Orthop Sports Phys Ther. 2017 Mar;47(3):180-189. doi: 10.2519/jospt.2017.7003. Epub 2016 Nov 5. PMID 27817301
- [Background] Bodkin SG, Bruce AS, Hertel J, Diduch DR, Saliba SA, Novicoff WM, Hart JM. Visuomotor therapy modulates corticospinal excitability in patients following anterior cruciate ligament reconstruction: A randomized crossover trial. Clin Biomech (Bristol). 2021 Jan;81:105238. doi: 10.1016/j.clinbiomech.2020.105238. Epub 2020 Nov 20. PMID 33234323
- [Background] Moraiti CO, Stergiou N, Vasiliadis HS, Motsis E, Georgoulis A. Anterior cruciate ligament reconstruction results in alterations in gait variability. Gait Posture. 2010 Jun;32(2):169-75. doi: 10.1016/j.gaitpost.2010.04.008. Epub 2010 Jun 29. PMID 20591671
- [Background] Vaz JR, Groff BR, Rowen DA, Knarr BA, Stergiou N. Synchronization dynamics modulates stride-to-stride fluctuations when walking to an invariant but not to a fractal-like stimulus. Neurosci Lett. 2019 Jun 21;704:28-35. doi: 10.1016/j.neulet.2019.03.040. Epub 2019 Mar 25. PMID 30922850
- [Background] Vaz JR, Knarr BA, Stergiou N. Gait complexity is acutely restored in older adults when walking to a fractal-like visual stimulus. Hum Mov Sci. 2020 Dec;74:102677. doi: 10.1016/j.humov.2020.102677. Epub 2020 Oct 15. PMID 33069099